CLINICAL TRIAL: NCT05326737
Title: Evaluation of Pain Trajectories After Surgery and Their Potential Relationship With Chronicity at 3 Months: a Single-center Prospective Cohort Study
Brief Title: Evaluation of Pain Trajectories After Surgery and Their Potential Relationship With Chronicity at 3 Months
Acronym: ETADOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2020/PC-02; 2020-A03223-36 (Other: RCB number)
Record Dates: First submitted 2022-04-04; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Surgical Procedures, Operative; Pain; Chronic Pain
Keywords: pain trajectory
MeSH Terms: conditions — Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population: The study population consists of adult surgery patients at the Nîmes University Hospital, with recruitment based on the operating theater program and for a predefined list of surgeries.
  Interventions: Other: In hospital pain evaluation; Other: In hospital questionnaires; Other: Telephone contact at 3 months

INTERVENTIONS:
Other: In hospital pain evaluation — Patients will evaluate their pain levels via a verbal numerical scale on days 1(or-1), 2, 3, 4, 5, 6 & 7.
Other: In hospital questionnaires — Patients are required to fill out the PCS questionnaire between on day -1 or +1.
Other: Telephone contact at 3 months — Patients will be contacted at 3 months post-surgery for pain questionnaires DN4 and EQ5D5L.

SUMMARY:
The effective management of acute postoperative pain remains a daily challenge despite the organizational efforts made and the techniques put in place.

Thirty percent of patients who undergo surgery suffer from chronic post-surgical pain, of which 5 to 10% are of severe intensity. Many preoperative, intraoperative, and postoperative factors, related to the patient, the surgical procedure, or the anesthetic technique, have been incriminated as risk factors for chronic post-surgical pain. The severity of acute postoperative pain is recognized as one of the risk factors for the occurrence of chronic post-surgical pain on which we can hope to interact during the peri-operative period.

In this cohort study, we wish to define the typologies of postoperative pain trajectories observed from Day 0 to Day 7 and to estimate the proportion of patients with an abnormal resolution of pain in a model of organization such as that of our institution, in classic hospitalization and in ambulatory care.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 3 months of follow-up
* The patient has undergone a planned surgical procedure in one of the participating departments
* The patient is willing and able to respond to the study questionnaires

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* It is impossible to correctly inform the patient
* Patient admitted to the ICU and still intubated at day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult surgery patients at the Nîmes University Hospital, with recruitment based on the operating theater program ffor a predefined list of surgeries.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-02-23 (Estimated); Study Completion 2024-05-23 (Estimated)

PRIMARY OUTCOMES:
The pain trajectory for the first 7 post-operative days. | Day 7
  The pain trajectory is the change in pain level evaluated by verbal numerical pain (from 0 to 10) from day 0 (surgery) to day 7.

SECONDARY OUTCOMES:
The DN4 questionnaire | month 3
  The Douleur Neuropathique 4 (DN4) questionnaire was developed by the French Neuropathic Pain Group and is a simple and objective tool, with the ability to distinguish nociceptive from neuropathic pain
The EuroQuol EQ5D5L questionnaire | month 3
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Since the surgery, do you have persistent pain? yes/no | month 3
  Since the surgery, do you have persistent pain? yes/no
Verbal numerical scale for pain (ranging from 0 to 10) | month 3
  Verbal numerical scale for pain (ranging from 0 to 10)
Have you had complications from your surgery? yes/no | month 3
  Have you had complications from your surgery? yes/no
Pain Catastrophizing Scale (PCS) | day -1 or day +1
  The Pain Catastrophizing Scale (PCS) is a 13-item self-report measure designed to assess catastrophic thinking related to pain among adults with or without chronic pain.
Cumulative consumption of antalgic drugs | day -1 or day +1
  Cumulative consumption of antalgic drugs
Cumulative consumption of antalgic drugs | day 2
  Cumulative consumption of antalgic drugs
Cumulative consumption of antalgic drugs | day 3
  Cumulative consumption of antalgic drugs
Cumulative consumption of antalgic drugs | day 4
  Cumulative consumption of antalgic drugs
Cumulative consumption of antalgic drugs | day 5
  Cumulative consumption of antalgic drugs
Cumulative consumption of antalgic drugs | day 6
  Cumulative consumption of antalgic drugs
Cumulative consumption of antalgic drugs | day 7
  Cumulative consumption of antalgic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Joël L'Hermite, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Background] Bouhassira D, Attal N, Alchaar H, Boureau F, Brochet B, Bruxelle J, Cunin G, Fermanian J, Ginies P, Grun-Overdyking A, Jafari-Schluep H, Lanteri-Minet M, Laurent B, Mick G, Serrie A, Valade D, Vicaut E. Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain. 2005 Mar;114(1-2):29-36. doi: 10.1016/j.pain.2004.12.010. Epub 2005 Jan 26. PMID 15733628
- [Background] Sullivan, M. J., Bishop, S. R., & Pivik, J. The pain catastrophizing scale: development and validation. Psychological assessment, 1995, 7(4), 524.